CLINICAL TRIAL: NCT00206297
Title: The Effect of Prolonged Pramlintide Infusion in Pediatric Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sponsored Programs, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-14358
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; hypoglycemia; hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia | interventions — pramlintide

INTERVENTIONS:
Drug: Pramlintide

SUMMARY:
The purpose of this study is to see if reducing the dose of insulin before a meal and giving both pramlintide and insulin as dual wave infusions will lower the chance of low blood sugars after a meal. In addition, the study will look at giving pramlintide as a basal infusion (a very low steady dose) for several hours

DETAILED DESCRIPTION:
The Diabetes Control and Complications Trial (DCCT) showed that improving blood sugar control for individuals with Type 1 diabetes (T1DM) stopped or delayed the onset of long-term complications. As a result of the study, intensive insulin management is aimed to control blood sugar and glycosylated hemoglobin (3 month blood glucose average test) as near to normal as safely possible. However, hypoglycemia (low blood sugar) was increased three fold in the DCCT study and is the major limiting factor in gaining "tight" control of blood sugar in T1DM.

In healthy individuals, an "after meal" blood sugar level is very carefully controlled. Insulin (the hormone that lowers blood sugar) and glucagon (hormone that raises blood sugar) play a key role in maintaining this careful balance. In T1DM, there is a lack of insulin and failure of glucagon suppression (keeping glucagon from being made too much). This leads to hyperglycemia (high blood sugar) right after you eat food. Also, glucagon is not controlled correctly after a meal. The glucagon, normally produced by the body, does not increase when a person with T1DM has a low blood sugar. This interferes with the balance between how much glucose is made and how much glucose is used. Therefore, glucagon fails to protect against low blood sugar in people with T1DM. This makes it very difficult to have normal blood sugars when someone has T1DM. This imbalance may be due to another hormone called amylin. This hormone may be too low in people with T1DM.

Amylin is produced in the pancreas (the part of the body that makes insulin) by the same cells that produce insulin and is also lacking in persons with T1DM. Amylin works by lowering glucagon after a meal. This keeps the liver from letting out stored sugar into the blood stream right after we eat. Pramlintide is man-made amylin and is given as a subcutaneous shot (under the skin) similar to insulin. At present, pramlintide has not received FDA approval.

Studies performed in adults have shown that adding amylin in T1DM, using pramlintide, lowers the high levels of glucagon made after a meal. This results in improved "after meal" high blood sugars and overall blood sugar control. Currently, pramlintide in adults is given as a separate injection from insulin, before meals, three times a day. When given as a bolus shot (one dose shot given all at once) to children and young adults, it seems to cause immediate low blood sugars after a meal. The low blood sugars may be caused by the "slowing down" of food digestion by pramlintide. Another possible cause of the low blood sugars may be the way pramlintide is being given (bolus shot versus a dual wave infusion).

ELIGIBILITY:
Inclusion Criteria:

Twenty (20) children with T1DM will be recruited for these studies. These children will be subjects of the Texas Children's Hospital Diabetes Care Center. The subjects must be:

1. Between 12-21 years of age at the time of enrollment.
2. Have been diagnosed with diabetes for at least 2 years and in good control (HbA1C less than 8.5%).
3. Be on continuous subcutaneous insulin infusion using an insulin pump.
4. Subjects must be otherwise healthy except for their T1DM and treated hypothyroidism.
5. Menstruating women must have a negative pregnancy test.
6. Hemoglobin equal to or > 12 g/dL before each study.
7. Weight more than 44 kg. -

Exclusion Criteria:

1. Age greater than 22 years or less than 12 years at the time of study
2. Any chronic disease: leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis, etc or on treatment that might directly or indirectly affect glucose homeostasis, except for diabetes and hypothyroidism stable on medications
3. Anemia (hemoglobin less than 12mg/dl)
4. Lack of a supportive family environment
5. Positive pregnancy test in menstruating young women
6. Evidence or history of chemical abuse
7. Hgb A1C greater than or equal to 8.5 % in a diabetic subject
8. BMI > 90 % tile for age or < 10 % tile for age
9. Weight less than 44 kg. -

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2003-10; Study Completion 2006-02

PRIMARY OUTCOMES:
Area under the curve for glucose

SECONDARY OUTCOMES:
glucagon and gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States